CLINICAL TRIAL: NCT03196505
Title: The Effect of Liposomal Bupivacaine on Post Operative Pain and Narcotic Use After Bariatric Surgery
Acronym: Exparel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017061
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Results first posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Bariatric Surgery Candidate; Pain, Postoperative
Keywords: Anesthetics, Local; Liposomal Bupivacaine; Bupivacaine; Postoperative Complications; Roux-en-Y Gastric Bypass; Sleeve Gastrectomy; Laparoscopic Bariatric Surgery
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications | interventions — Injections; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Liposomal Bupivacaine (Active Comparator): Liposomal bupivacaine (Exparel) 20mL of injectable saline diluted with 60 ml of 0.25% Marcaine and 20 ml of saline for a total of 100 ml. After induction of anesthesia, the patients will receive a 20 ml mixture locally infiltrated at each trocar incision site (5 sites).
  Interventions: Drug: Exparel 266 MG Per 20 ML Injection
- Control (Active Comparator): 60 milliliters (ml) of 0.25% bupivacaine diluted with 40 ml of saline for a total of 100 ml. After induction of anesthesia, the patients will receive 20 ml mixture locally infiltrated at each trocar incision site (5 sites).
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Exparel 266 MG Per 20 ML Injection — Liposomal bupivacaine 20mL of injectable saline diluted with 60 ml of 0.25% Marcaine and 20 ml of saline for a total of 100 ml. After induction of anesthesia, the patients will receive a 20 ml mixture locally infiltrated at each trocar incision site (5 sites).
  Other Names: EXPAREL
  Arms: Liposomal Bupivacaine
Drug: Bupivacaine — 60 milliliters (ml) of 0.25% bupivacaine diluted with 40 ml of saline for a total of 100 ml. After induction of anesthesia, the patients will receive 20 ml mixture locally infiltrated at each trocar incision site (5 sites).
  Other Names: Marcaine
  Arms: Control

SUMMARY:
This study is prospective, randomized trial in which the efficacy of liposomal bupivacaine (Exparel®) is compared to standard bupivacaine local surgical site injection in reducing total IV and oral morphine equivalents required after laparoscopic bariatric surgery. Liposomal bupivacaine is a 72-hour bupivacaine that is slowly released from tissue over the course of three days. Having a long acting local anesthetic should provide better pain control than conventional bupivacaine which has a 3.5-hour half-life. In some studies, the use of liposomal bupivacaine has been shown to decrease pain and narcotic use after surgery. This has not yet been studied in bariatric patients and the use of liposomal bupivacaine can potentially improve patient post-operative pain control, decrease narcotic use, decrease hospital length of stay and readmission rates and improve patient satisfaction after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing elective laparoscopic sleeve gastrectomy or Roux-en-Y gastric bypass surgeries.
* Fulfills NIH criteria for bariatric surgery

Exclusion Criteria:

* Patients deemed not a candidate for laparoscopic bariatric surgery
* Patients with previous bariatric or gastric surgeries.
* BMI <35 and > 60 kg/m2
* Preoperative inability to ambulate and confined to wheelchair.
* American Society of Anesthesiologist (ASA) score >3
* Concurrent ventral hernia repair or intraoperative extensive lysis of adhesions
* Not able to understand informed consent, or unwilling to sign consent.
* Not able to understand and read English
* Currently pregnant or lactating.
* Age <18 or >65
* Patients intolerant of opiates, NSAIDS, acetaminophen or local anesthetics.
* Patients requiring opiate use within 30 days prior to time of surgery.
* Patients with reported use of narcotics greater than 2 weeks in preceding year before surgery.
* Patients with history of substance abuse, alcohol addiction
* Patients with diagnosis of chronic pain, history of fibromyalgia, chronic regional pain syndrome (dystrophic pain syndrome).
* Bupivacaine use within 96 hours before operation
* Prisoners
* Bariatric surgery operation >3 hours.
* More than 5 laparoscopic incision sites used during surgery, conversion to open operation, placement of a feeding tube or drain.
* Patients with renal failure or hepatic failure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pearl Ma, MD, Principal Investigator — University of San Francisco - Fresno
Locations (1):
- Fresno Heart and Surgical Hospital, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ma P, Lloyd A, McGrath M, Shuchleib Cung A, Akusoba I, Jackson A, Swartz D, Boone K, Higa K. Efficacy of liposomal bupivacaine versus bupivacaine in port site injections on postoperative pain within enhanced recovery after bariatric surgery program: a randomized clinical trial. Surg Obes Relat Dis. 2019 Sep;15(9):1554-1562. doi: 10.1016/j.soard.2019.06.004. Epub 2019 Jun 17. PMID 31375443

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liposomal Bupivacaine | Control
Started | 115 | 116
Completed | 89 | 90
Not Completed | 26 | 26
Not completed — Physician Decision | 26 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liposomal Bupivacaine | Control | Total
Number analyzed (Participants) | 89 | 90 | 179
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 89 | 90 | 179
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (9.8) | 39.2 (10.1) | 39.2 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 74 | 142
  Male | 21 | 16 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] — BMI is Calculated as Kg/m^2
  Kg/m^2 | 45.4 (5.9) | 44.5 (5.5) | 45 (5.7)
Diabetes [Count of Participants; unit: Participants] | 13 | 13 | 26
Hypertension [Count of Participants; unit: Participants] | 35 | 29 | 64

OUTCOME MEASURES:

1. Primary Outcome: Morphine Equivalents
Description: in hospital total oral and IV morphine equivalents required after laparoscopic bariatric surgery.
Time Frame: within 1 week post-operatively
Measure: Mean (Standard Deviation); unit: MEU
Arm/Group | Liposomal Bupivacaine | Control
Number analyzed (Participants) | 89 | 90
MEU | 8.3 (4.0) | 7.5 (3.6)

2. Secondary Outcome: Cumulative Pain Score
Description: Average pain scores by blinded nurse obtained. Analogue pain rating scale ranged from 0 to 10 with 0 being no pain and 10 being the worst possible pain. Assessment of pain and nausea were performed every 4 hours after operation until discharge.
Time Frame: within 48 hours post operatively
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Liposomal Bupivacaine | Control
Number analyzed (Participants) | 89 | 90
score on a scale | 3.5 (1.7) | 3.6 (1.9)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Liposomal Bupivacaine | Control
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/90
Serious Adverse Events (participants affected / at risk) | 5/89 | 3/90
Other Adverse Events (participants affected / at risk) | 0/89 | 0/90
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liposomal Bupivacaine (N=89) | Control (N=90)
Readmission to hospital (Gastrointestinal disorders) | 3 (3) | 3 (3) — Nausea requiring IV hydration
Reoperations (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Bleeding

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT03196505/Prot_SAP_000.pdf